CLINICAL TRIAL: NCT05305248
Title: Comparison of Sedation With Intravenous Remimazolam and Dexmedetomidine During Spinal Anesthesia : Prospective Randomized Study
Brief Title: Sedation With Remimazolam During Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Do-Hyeong Kim, Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3-2021-0489
Record Dates: First submitted 2022-03-02; First posted 2022-03-31 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Sedation; Spinal Anesthesia
MeSH Terms: interventions — remimazolam; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam group (Experimental): Sedation with remimazolam during spinal anesthesia
  Interventions: Drug: Remimazolam
- Dexmedetomidine group (Active Comparator): Sedation with dexmedetomidine during spinal anesthesia
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Remimazolam — After spinal anesthesia, 5 mg of remimazolam is injected by intravenous route for 1 minute to induce sedation. To maintain sedation, remimazolam is continuously infused at a rate within the range of 0.1 mg/kg/h to 1 mg/kg/h.
  Arms: Remimazolam group
Drug: Dexmedetomidine — After performing spinal anesthesia, dexmedetomidine is injected at a loading dose of 1 mcg/kg for 10 minutes to induce sedation. Thereafter, to maintain sedation, Dexmedetomidine is continuously infused at a rate within the range of 0.2 to 0.7 mcg/kg/h.
  Arms: Dexmedetomidine group

SUMMARY:
Remimazolam is a benzodiazepine-binding site antagonist of the GABA receptor, metabolized by esterases, and exhibits a stable context-sensitive half-life of 6-7 minutes. Remimazolam has a high clearance rate and a small volume of distribution in the pharmacokinetic model. The US FDA has approved sedation for surgery. Although there have been studies on the use of remimazolam as a sedative for procedures such as endoscopy, there have been no reports of the use of remimazolam in spinal anesthesia. The purpose of this study is to compare and analyze the hemodynamics and recovery profile of patients undergoing surgery under spinal anesthesia by maintaining sedation with dexmedetomidine or remimazolam.

ELIGIBILITY:
Inclusion Criteria:

1. Severe cardiovascular or respiratory disease
2. Contraindication to spinal anesthesia
3. Heart block
4. Previous hepatectomy or liver transplant
5. Patients with moderate or more hepatic impairment (AST/ALT is more than 2.5 times the upper limit of normal)
6. Estimated glomerular filtration rate < 30 mL/min/1.73m2
7. Acute narrow angle glaucoma
8. Myasthesia gravis
9. Known allergy to the drugs included in the study

Exclusion Criteria:

1. Patients 19 years of age or older who are expected to elective orthopedic surgery under spinal anaesthesia
2. ASA PS 1-3

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
MOAA/S score | up to 30 minutes after PACU arrival
  MOAA/S score will be evaluated by an 5-point scale from iniation of sedative drugs to 30 minutes after PCAU arrival at 10 minutes intervals.

SECONDARY OUTCOMES:
Sedation induction time Sedation induction time | up to 5 minutes after initation of sedative drugs
  Sedation induction time is defined as from start of drug injection to the first time of MOAA/S ≤ 3
Differences in basic vital signs between the two groups | Baseline
  Differences in blood pressure, heart rate, and patient sedation index at different time points during the operation and PACU stay between the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No